CLINICAL TRIAL: NCT02172066
Title: Evaluation of the Narrative Exposure Therapy (NET) as Means to Reduce Psychological Impairment in the Aftermath of the Recent Flood Disaster in Bujumbura, Burundi
Brief Title: Narrative Exposure Therapy (NET) for Victims of the Recent Flood Disaster in Burundi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Vivo international e.V. (Industry); Université Lumière de Bujumbura (Other)
Responsible Party: Principal Investigator, Anselm Crombach, Principal Investigator, University of Konstanz
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UKCR2014
Record Dates: First submitted 2014-06-19; First posted 2014-06-24 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Childhood maltreatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Narrative Exposure Therapy (NET) (Experimental): During NET, the client, with the assistance of the therapist, constructs a chronological narrative of his or her entire life with a focus on exposure to traumatic stress. Empathic understanding, active listening, congruency and unconditional positive regard are key components of the therapist's behavior. The therapist asks in detail for emotions, cognitions, sensory information, and physiological reactions to link the traumatic events to an autobiographical context, namely time and place. In total the Individuals receive 6 sessions of NET, every session lasting between 1,5 and 2 hr depending on the needs of the participant.
  Interventions: Behavioral: Narrative Exposure Therapy (NET)
- No treatment control (No Intervention)

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy (NET)
  Arms: Narrative Exposure Therapy (NET)

SUMMARY:
In the aftermath of natural disasters, e.g., flood disasters, there is a great need for humanitarian assistance in the domain of psychological support. This is particularly true in post-conflict settings because people have suffered severely from multiple traumatic events and situations during their lives. The Narrative Exposure Therapy (NET) is a short-term, culturally sensitive treatment approach that aims to reduce Posttraumatic Stress Disorder (PTSD) symptoms.

The investigators want to provide evidence, that NET is an effective and efficient module to assist people in the aftermath of natural disasters using the example of the recent flood disaster in Burundi. In addition the investigators aim to explore, how traumatic incidences and maltreatment during childhood may influence treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals severely affected (e.g., who had lost their children) by the flood disaster in Bujumbura
* All participants were part of the emergency program of the Red Cross Burundi who assisted those most affected by the flood disaster in Bujumbura
* Inclusion criteria for therapy: High degree of symptoms of posttraumatic stress disorder according to the Posttraumatic Symptom Scale - Interview (PSSI)

Exclusion Criteria:

* Pregnancy
* Current substance dependence
* Psychotic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Diagnosis and load of PTSD symptoms assessed via the Posttraumatic Symptom Scale - Interview (PSS-I) at 3 and 9 months follow-up | baseline, 3-months-follow-up, 9-months-follow-up

SECONDARY OUTCOMES:
Change from baseline in load of depressive symptoms assessed via the Patient Health Questionnaire-9 (PHQ-9) at 3 months and 9 months follow-up | baseline, 3-months-follow-up, 9-months-follow-up
Change in strength of suicidal ideation measured via the Mini International Neuropsychiatric Interview (M.I.N.I.) at 3 months and 6 months follow-up | baseline, 3-months-follow-up, 9-months-follow-up

OTHER OUTCOMES:
Previous traumatic events measured via vivo Event Checklist for War, Detention and Torture Experiences | baseline
Adverse experiences during childhood measured via the Domestic and Community Violence Checklist | 3-months-follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Anselm Crombach, Dr, Principal Investigator — University of Konstanz
Locations (1):
- vivo international e.V.; University Lumière de Bujumbura; Red Cross Burundi, Bujumbura, Burundi